CLINICAL TRIAL: NCT01083719
Title: Phase II Study Comparing FDG-PET Versus MRI Based Target Volume Delineation in Glioblastoma and the Role of FDG-PET/CT in the Alteration of MRI Based Target Volumes.
Brief Title: A Comparison of FDG-PET Versus MRI Based Target Volume Delineation in Glioblastoma and the Role of FDG-PET/CT in the Alteration of MRI Based Target Volumes.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medanta Institute of Clinical Research (Other)
Responsible Party: Dr. Tejinder kataria/ principal Investigator, Medanta- The medicity
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AHD1234
Record Dates: First submitted 2010-03-06; First posted 2010-03-10 (Estimated); Last update posted 2010-03-10 (Estimated); Status verified 2010-03

CONDITIONS: Glioblastoma
Keywords: Glioblastoma; FDG-PET; MRI
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FDG-PET (Experimental): A comparison of FDG-PET versus MRI based target volume delineation in glioblastoma and the role of FDG-PET/CT in the alteration of MRI based target volumes.
  Interventions: Procedure: FDG-PET

INTERVENTIONS:
Procedure: FDG-PET — Fluoro-deoxy gluocose-Positron emission tomography for delineating volumes in Glioblastoma

SUMMARY:
HYPOTHESIS AND SAMPLE SIZE The tumor delineated by FDG-PET is significantly different from the delineation achieved by MR T1 contrast weighted images in glioblastoma; expecting a standard error of 12.5 % (a confidence interval of 25%), with a confidence level set at 95%, a sample size of 15 patients would be accrued in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Post operative patients of documented high grade gliomas (grade III and IV)
2. Patients who have not undergone any previous irradiation to brain.
3. Performance Scale as defined by ECOG PS 0-3

Exclusion Criteria:

1. Patients who are diabetic.
2. Patients who are pregnant.
3. Any documented contrast allergy to the agents used for imaging.
4. Patients who are unable to comprehend or cooperate effectively for treatment planning.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-08 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
Tumor infiltration defined on FDG-PET not determined to MRI | 18 months